CLINICAL TRIAL: NCT04940143
Title: The Evaluation of Effects of Botulinum Toxin Injection on Lower Extremity Somatosensory Impairment and Postural Control in Children With Hemiplegic Cerebral Palsy
Brief Title: Effects of Botulinum Toxin Injection on Sensation and Postural Control in Children With Hemiplegic Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09.2020.863
Record Dates: First submitted 2021-06-17; First posted 2021-06-25 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Cerebral Palsy; Hemiplegic Cerebral Palsy
Keywords: Botulinum toxin; Hemiplegic cerebral palsy; Postural control; Sensory function; Balance
MeSH Terms: conditions — Cerebral Palsy | interventions — Botulinum Toxins, Type A; Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Botulinum toxin-A (Experimental): Botulinum toxin-A (Onabotulinum toxin type-A) injection with electrical stimulation guidance will be administered to spastic ankle plantar flexor muscles. After the injection, the patients will be included in the comprehensive physiotherapy program.
  Interventions: Drug: Botulinum toxin type-A (Onabotulinum toxin type-A); Other: Physical Therapy

INTERVENTIONS:
Drug: Botulinum toxin type-A (Onabotulinum toxin type-A) — Botulinum toxin-A (Onabotulinum toxin type-A/Botox®) injection will be administered from three different points, two on the medial head of the gastrocnemius muscle and one point on the lateral head with total 3-6 units/kg dose, under the guidance of electrical stimulation for the detection of the target neuromuscular junction.
Other: Physical Therapy — After the botulinum toxin-A injection, the patients will be included in the comprehensive physiotherapy program thrice a week for a total of 12 weeks. The physiotherapy program will be consisted of the ankle range of motion and stretching, strengthening of the antagonist muscles, proprioception exercises, functional walking training and static and dynamic balance training.

SUMMARY:
In this study, the investigators aimed to investigate the effects of botulinum neurotoxin type A (BoNT-A) injection applied to the ankle plantar flexor muscles on lower extremity sensation and quantitative balance parameters in children with spastic hemiplegic cerebral palsy who are ambulatory without an assistive device in daily life.

DETAILED DESCRIPTION:
Cerebral palsy (CP) refers to a group of movement and posture disorders that limit activity and participation, that are attributed to non-progressive disturbances in the developing fetus or infant brain. One of the main clinical findings of CP is postural control disorder. Many concomitant impairments such as joint range of motion limitations, spasticity, contractures, sensory deficits and loss of selective motor control contribute to postural control disorder.

One of the most common causes of motor dysfunction in children with CP is the presence of spasticity. Spasticity in the ankle plantar flexor muscles and weakness in the dorsiflexor muscles are the main factors that cause gait disturbance. Thus, impairments in gait function cause limitation of postural stability. Although there are many methods in spasticity management, BoNT-A injections have been used effectively and safely for many years, especially in reducing ankle plantar flexor spasticity. There are limited number of studies in the literature investigating the effect of BoNT-A injection on postural control in children with spastic CP, and only one study included children with spastic hemiplegic (unilateral) CP and it was clearly highlighted that new studies are needed in this area.

The reclassification of CP acknowledges the contribution of impaired sensation in motor performance. Although it has been shown that somatosensory deficits in the lower extremities of children with spastic CP can negatively affect gait and balance, the effect of spasticity in the ankle has not been evaluated.

In this study, the investigators aimed to investigate the effects of BoNT injection applied to the ankle plantar flexor muscles on lower extremity sensation and quantitative balance parameters in children with spastic hemiplegic CP who are ambulatory without an assistive device in daily life.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with hemiplegic cerebral palsy
* Age between 5-13 years
* MAS ≥ 2 spasticity in the affected ankle
* Gross Motor Function Classification System (GMFCS) level I-II
* Able to understand given commands
* Sufficient cooperation to understand instructions and participate evaluations
* Giving an informed consent
* Botulinum toxin A injection decision made by an experienced Physiatrist

Exclusion Criteria:

* Visual, vestibular and cognitive deficits
* Botulinum toxin A treatment within 6 months or having undergone an orthopaedic surgery 1 year prior to inclusion in the study
* Presence of fixed contracture or joint instability in the affected ankle
* Severe scoliosis (Cobb angle >40°)
* Uncontrolled epilepsy
* Having undergone selective dorsal rhizotomy

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 19 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Modified Clinical Test of Sensory Interaction on Balance (mCTSIB) of NeuroCom Balance Master | before intervention (T0)
  Modified Clinical Test of Sensory Interaction on Balance (mCTSIB) will be done by Balance Master device. Postural sway velocities (degree/second) will be recorded on the firm and foam surfaces with eyes opened and closed conditions of mCTSIB test. Higher scores mean worse static postural stability.
Modified Clinical Test of Sensory Interaction on Balance (mCTSIB) test of NeuroCom Balance Master | 4th week after intervention (T1)
  Modified Clinical Test of Sensory Interaction on Balance (mCTSIB) test will be done by Balance Master device. Postural sway velocities (degree/second) will be recorded on the firm and foam surfaces with eyes opened and closed conditions of mCTSIB test. Higher scores mean worse static postural stability.
Modified Clinical Test of Sensory Interaction on Balance (mCTSIB) test of NeuroCom Balance Master | 3rd month after intervention (T2)
  Modified Clinical Test of Sensory Interaction on Balance (mCTSIB) test will be done by Balance Master device. Postural sway velocities (degree/second) will be recorded on the firm and foam surfaces with eyes opened and closed conditions of mCTSIB test. Higher scores mean worse static postural stability.
Light touch pressure treshold | before intervention (T0)
  Light touch pressure (tactile) sensation will be assessed by using Semmes-Weinstein Monofilaments kit (Baseline, White Plains, New York, NY,USA) at the first and fifth metatarsal heads and heel of the plantar side of each foot. The light touch pressure threshold will be defined as the thinner monofilament value the participant correctly identified twice out of three trials for each application site. Higher scores mean worse tactile sensation.
Light touch pressure treshold | 4th week after intervention (T1)
  Light touch pressure (tactile) sensation will be assessed by using Semmes-Weinstein Monofilaments kit (Baseline, White Plains, New York, NY,USA) at the first and fifth metatarsal heads and heel of the plantar side of each foot. The light touch pressure threshold will be defined as the thinner monofilament value the participant correctly identified twice out of three trials for each application site. Higher scores mean worse tactile sensation.
Light touch pressure treshold | 3rd month after intervention (T2)
  Light touch pressure (tactile) sensation will be assessed by using Semmes-Weinstein Monofilaments kit (Baseline, White Plains, New York, NY,USA) at the first and fifth metatarsal heads and heel of the plantar side of each foot. The light touch pressure threshold will be defined as the thinner monofilament value the participant correctly identified twice out of three trials for each application site. Higher scores mean worse tactile sensation.

SECONDARY OUTCOMES:
Modified Ashworth Scale (MAS) | before intervention (T0)
  Muscle tone and spasticity will be measured with MAS. Muscle tone is scored between 0-4. Higher scores mean more severe spasticity.
Modified Ashworth Scale (MAS) | 4th week after intervention (T1)
  Muscle tone and spasticity will be measured with MAS. Muscle tone is scored between 0-4. Higher scores mean more severe spasticity.
Modified Ashworth Scale (MAS) | 3rd month after intervention (T2)
  Muscle tone and spasticity will be measured with MAS. Muscle tone is scored between 0-4. Higher scores mean more severe spasticity.
Modified Tardieu Scale (MTS) | before intervention (T0)
  Within the Modified Tardieu Scale (MTS), angle of arrest of the ankle joint at slow speed (XV1), angle of catch at fast speed (XV3), spasticity grade (Y), and spasticity angle (X) will be recorded. Angles of arrest and catch will be measured by a goniometer and angle of arrest of the ankle joint at slow speed was recorded as passive range of motion. Higher X angle points out dynamic component of spasticity. Higher Y scores mean more severe spasticity.
Modified Tardieu Scale (MTS) | 4th week after intervention (T1)
  Within the Modified Tardieu Scale (MTS), angle of arrest of the ankle joint at slow speed (XV1), angle of catch at fast speed (XV3), spasticity grade (Y), and spasticity angle (X) will be recorded. Angles of arrest and catch will be measured by a goniometer and angle of arrest of the ankle joint at slow speed was recorded as passive range of motion. Higher X angle points out dynamic component of spasticity. Higher Y scores mean more severe spasticity.
Modified Tardieu Scale (MTS) | 3rd month after intervention (T2)
  Within the Modified Tardieu Scale (MTS), angle of arrest of the ankle joint at slow speed (XV1), angle of catch at fast speed (XV3), spasticity grade (Y), and spasticity angle (X) will be recorded. Angles of arrest and catch will be measured by a goniometer and angle of arrest of the ankle joint at slow speed was recorded as passive range of motion. Higher X angle points out dynamic component of spasticity. Higher Y scores mean more severe spasticity.
Sit to Stand (STS) test of Neurocom Balance Master | before intervention (T0)
  The Sit to stand (STS) test will be done by Balance Master device. Weight transfer time (sec), rising index (%) and sway velocity (deg/sec) will be recorded. The STS is a performance test quantifying the patient's ability, on command, to quickly rise from a seated to a standing position. The STS quantifies time required to transfer weight from the buttock to the feet (weight transfer time (sec)), the strength of the rise (rising index (%)), and the center of gravity sway velocity (deg/sec) during the rise to stand and the first five seconds during standing. Higher scores mean worse dynamic postural control.
Sit to Stand (STS) test of Neurocom Balance Master | 4th week after intervention (T1)
  The Sit to stand (STS) test will be done by Balance Master device. Weight transfer time (sec), rising index (%) and sway velocity (deg/sec) will be recorded. The STS is a performance test quantifying the patient's ability, on command, to quickly rise from a seated to a standing position. The STS quantifies time required to transfer weight from the buttock to the feet (weight transfer time (sec)), the strength of the rise (rising index (%)), and the center of gravity sway velocity (deg/sec) during the rise to stand and the first five seconds during standing. Higher scores mean worse dynamic postural control.
Sit to Stand (STS) test of Neurocom Balance Master | 3rd month after intervention (T2)
  The Sit to stand (STS) test will be done by Balance Master device. Weight transfer time (sec), rising index (%) and sway velocity (deg/sec) will be recorded. The STS is a performance test quantifying the patient's ability, on command, to quickly rise from a seated to a standing position. The STS quantifies time required to transfer weight from the buttock to the feet (weight transfer time (sec)), the strength of the rise (rising index (%)), and the center of gravity sway velocity (deg/sec) during the rise to stand and the first five seconds during standing. Higher scores mean worse dynamic postural control.
Step&Quick Turn (SQT) test of Neurocom Balance Master | before intervention (T0)
  The Step&Quick Turn (SQT) test will be done by Balance Master device. The SQT is a performance test that quantifies turn performance characteristics. The patient is instructed to take two forward steps on command, and then quickly turn 180˚ to either the left or right and return to the starting point. The time required to execute the turn (sec), and the velocity of COG sway (deg) during the turn will be recorded. Higher scores mean worse dynamic postural control.
Step&Quick Turn (SQT) test of Neurocom Balance Master | 4th week after intervention (T1)
  The Step&Quick Turn (SQT) test will be done by Balance Master device. The SQT is a performance test that quantifies turn performance characteristics. The patient is instructed to take two forward steps on command, and then quickly turn 180˚ to either the left or right and return to the starting point. The time required to execute the turn (sec), and the velocity of COG sway (deg) during the turn will be recorded. Higher scores mean worse dynamic postural control.
Step&Quick Turn (SQT) test of Neurocom Balance Master | 3rd month after intervention (T2)
  The Step&Quick Turn (SQT) test will be done by Balance Master device. The SQT is a performance test that quantifies turn performance characteristics. The patient is instructed to take two forward steps on command, and then quickly turn 180˚ to either the left or right and return to the starting point. The time required to execute the turn (sec), and the velocity of COG sway (deg) during the turn will be recorded. Higher scores mean worse dynamic postural control.
Two-point discrimination | before intervention (T0)
  Two-point discrimination will be assessed by using a discriminator (Baseline®, White Plains, New York, NY, USA) on the forefoot and heel of the plantar side of each foot, and scored as the minimum distance in mm between two stimulus points, which were correctly identified as distinct points twice out of three trials for each site. Higher scores mean worse two-point discrimination.
Two-point discrimination | 4th week after intervention (T1)
  Two-point discrimination will be assessed by using a discriminator (Baseline®, White Plains, New York, NY, USA) on the forefoot and heel of the plantar side of each foot, and scored as the minimum distance in mm between two stimulus points, which were correctly identified as distinct points twice out of three trials for each site. Higher scores mean worse two-point discrimination.
Two-point discrimination | 3rd month after intervention (T2)
  Two-point discrimination will be assessed by using a discriminator (Baseline®, White Plains, New York, NY, USA) on the forefoot and heel of the plantar side of each foot, and scored as the minimum distance in mm between two stimulus points, which were correctly identified as distinct points twice out of three trials for each site. Higher scores mean worse two-point discrimination.
Selective Control Assessment of the Lower Extremity (SCALE) | before intervention (T0)
  The lower extremity selective voluntary motor control will be assessed with SCALE tool. Hip, knee, ankle, subtalar, and toe joints are assessed bilaterally in SCALE. Selective voluntary motor control is graded at each joint as 'normal' (2 points), 'impaired' (1 point), or 'unable' (0 points). The SCALE score is the sum of each joint scores and assumes a 10 point maximum per limb. The total SCALE score is between 0-20 and higher scores mean better selective motor control.
Selective Control Assessment of the Lower Extremity (SCALE) | 4th week after intervention (T1)
  The lower extremity selective voluntary motor control will be assessed with SCALE tool. Hip, knee, ankle, subtalar, and toe joints are assessed bilaterally in SCALE. Selective voluntary motor control is graded at each joint as 'normal' (2 points), 'impaired' (1 point), or 'unable' (0 points). The SCALE score is the sum of each joint scores and assumes a 10 point maximum per limb. The total SCALE score is between 0-20 and higher scores mean better selective motor control.
Selective Control Assessment of the Lower Extremity (SCALE) | 3rd month after intervention (T2)
  The lower extremity selective voluntary motor control will be assessed with SCALE tool. Hip, knee, ankle, subtalar, and toe joints are assessed bilaterally in SCALE. Selective voluntary motor control is graded at each joint as 'normal' (2 points), 'impaired' (1 point), or 'unable' (0 points). The SCALE score is the sum of each joint scores and assumes a 10 point maximum per limb. The total SCALE score is between 0-20 and higher scores mean better selective motor control.
Timed Up and Go (TUG) test | before intervention (T0)
  Functional mobility and balance will be assessed the TUG test. It records the time a child needs to stand up from a chair with foot contact, to walk three meter to a target, turn around and return to the chair and sit down as quickly and safely as possible. The test will be repeated three times and the average time (sec) will be recorded. Higher scores mean worse functional mobility.
Timed Up and Go (TUG) test | 4th week after intervention (T1)
  Functional mobility and balance will be assessed the TUG test. It records the time a child needs to stand up from a chair with foot contact, to walk three meter to a target, turn around and return to the chair and sit down as quickly and safely as possible. The test will be repeated three times and the average time (sec) will be recorded. Higher scores mean worse functional mobility.
Timed Up and Go (TUG) test | 3rd month after intervention (T2)
  Functional mobility and balance will be assessed the TUG test. It records the time a child needs to stand up from a chair with foot contact, to walk three meter to a target, turn around and return to the chair and sit down as quickly and safely as possible. The test will be repeated three times and the average time (sec) will be recorded. Higher scores mean worse functional mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Evrim Karadag Saygi, Prof, Principal Investigator — Marmara University
Locations (1):
- Marmara University School of Medicine, Pendik Education and Research Hospital, Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No